CLINICAL TRIAL: NCT05420142
Title: Innovative plAnt Protein Fibre and Physical Activity Solutions to Address Poor appEtite and prevenT undernutrITion in oldEr Adults (APPETITE): Determination of In-vivo Plasma AA Appearance From Plant Protein Fibre Products
Brief Title: Determination of In-vivo Plasma AA Appearance From Plant Protein Fibre Products
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); University of Padova (Other); Fraunhofer Institute for Interfacial Engineering and Biotechnology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: APPETITE_AA3.1
Record Dates: First submitted 2022-05-04; First posted 2022-06-15 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Aging; Undernutrition; Appetite Loss; Age-Related Sarcopenia
Keywords: Amino Acid; Gut hormones; Older adults; Successful ageing; Plant protein; Fibre
MeSH Terms: conditions — Malnutrition; Anorexia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test meal incorporating the study groups innovative plant protein and fibre (variety 3) product. (Experimental): The standardised test meal was prepared in a single dose using Knorr low sodium chicken stock cubes (9g = 1 stock cube), 65.64g of plant protein and fibre variety 3 (3.09g leucine), 28.6g butter, 5.12g cornflour, and 300ml water. The test meal is consumed in a single sitting in the morning following an overnight fast. Blood samples are acquired at baseline and at set intervals over the subsequent 3-hours to examine the net peripheral amino acid appearance.
  Interventions: Dietary Supplement: Net peripheral AA appearance following ingestion of 3 selected PPF products compared to whey
- Test meal incorporating the study groups innovative plant protein and fibre (variety 5) product. (Experimental): The standardised test meal was prepared in a single dose using Knorr low sodium chicken stock cubes (9g = 1 stock cube), 67.78g of plant protein and fibre variety 3 (3.09g leucine), 27.79g butter, 4.63g cornflour, and 300ml water. The test meal is consumed in a single sitting in the morning following an overnight fast. Blood samples are acquired at baseline and at set intervals over the subsequent 3-hours to examine the net peripheral amino acid appearance.
  Interventions: Dietary Supplement: Net peripheral AA appearance following ingestion of 3 selected PPF products compared to whey
- Test meal incorporating the study groups innovative plant protein and fibre (variety 6) product. (Experimental): The standardised test meal was prepared in a single dose using Knorr low sodium chicken stock cubes (9g = 1 stock cube), 57.66g of plant protein and fibre variety 3 (3.09g leucine), 31.72g butter, 6.62g cornflour, and 300ml water. The test meal is consumed in a single sitting in the morning following an overnight fast. Blood samples are acquired at baseline and at set intervals over the subsequent 3-hours to examine the net peripheral amino acid appearance.
  Interventions: Dietary Supplement: Net peripheral AA appearance following ingestion of 3 selected PPF products compared to whey
- Test meal incorporating the control comparator (whey protein isolates), plus 10g of added pea fibre. (Active Comparator): The standardised test meal was prepared in a single dose using Knorr low sodium chicken stock cubes (9g = 1 stock cube), 36.59g of unflavoured Optimum Nutrition gold standard 100% whey protein (3.09g leucine), 33.23g butter, 9.09g cornflour, and 300ml water. The test meal is consumed in a single sitting in the morning following an overnight fast. Blood samples are acquired at baseline and at set intervals over the subsequent 3-hours to examine the net peripheral amino acid appearance.
  Interventions: Dietary Supplement: Net peripheral AA appearance following ingestion of 3 selected PPF products compared to whey

INTERVENTIONS:
Dietary Supplement: Net peripheral AA appearance following ingestion of 3 selected PPF products compared to whey — The intervention will assess the effects of three difference varieties of plant-based protein and fibre supplements on net peripheral amino acid appearance in blood compared to whey protein with matched fibre content as a control arm.

SUMMARY:
This study aims to assess the digestibility and efficacy of the study groups previously developed innovative plant-based protein and fibre products.

DETAILED DESCRIPTION:
Older people are at high risk of undernutrition, which leads to serious adverse health outcomes, but effective preventive strategies are lacking. Effective, new strategies should focus on the etiology of undernutrition and directly address potential causes and mechanisms underpinning undernutrition.

Reduced food intake and restricted dietary diversity are direct consequences of poor appetite. Recent studies have shown, that older persons with a poor appetite demonstrate lower intake of protein and dietary fibre, and of several nutrient-rich food groups (e.g. meat, fish, wholegrains, vegetables), after adjustment for energy intake and other potential confounders, but a higher consumption of food groups low in micronutrients (e.g. fats, oils, sweets, and sodas), compared to those with good appetite.

Enhancing dietary protein and fibre intake in older Europeans is a key objective because intake of both nutrients is sub- optimal, not only in those with poor appetite. Adequate protein intake prevents excessive decline in muscle mass and function (sarcopenia), a widespread health-issue in older persons, intensified by undernutrition. Adequate dietary fibre intake prevents constipation and impedes the development of many chronic diseases prevalent in older people. Thus, targeting adequate protein and fibre intake may be particularly beneficial in this vulnerable population.

A preparatory short-term study will be performed to assess in 10 healthy older adults the net peripheral Amino Acid (AA) appearance following ingestion of 3 selected Plant-based Proteins and Fibre (PPF) products previously developed by the wider study collaborators, compared to the reference of 30 g whey protein. Plasma concentrations of AA from arterialised blood will be measured by ion exchange chromatography in blood samples (1 drawn before and 6 during 3 hours postprandial). This step will allow the research group to compare in-vitro (previous work) and in-vivo digestibility of several PPF mixtures and identify the product with both optimal amino acid composition and sensory properties as well as optimal post-prandial plasma amino acid profile to be used in further studies.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling, Age 65+ years, not a heavy smoker (≤10/day), BMI 18-30 kg/m2

Exclusion Criteria:

* Medical condition or medication known to impact appetite or energy intake, consumes more than 14 (female) or 21 (male) units of alcohol per week, inability to come to study centre, self-reported cognitive impairment or diagnosis of clinical depression, heavy smoker (>10/day)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Acute change in amino acid appearance in peripheral blood following a test meal ingestion | Blood samples will be taken at baseline, and at 30, 60, 90, 120, 150, & 180 minutes following ingestion of test sample
  Arterialised blood samples will be drawn from antecubital vein and centrifuged at 4˚C for 10 minutes at 4000rpm and frozen at -80˚C until analysed. Samples will be analysed using HPLC methods and expressed in μmol/L.

SECONDARY OUTCOMES:
Acute changes in appetite and desire to eat | baseline, 30, 60, 90, 120, 150, & 180 minutes following ingestion of a sample meal
  Changes in appetite and are assessed at set time points throughout the testing session, matched for timing of biological sample collection. This will be assessed using the validated visual analogue scale (VAS) method. The Visual Analogue Scale is a 100mm scale with anchors on each end describing extreme answers. On the left side of the scale is the extreme negative response and the right side the positive response. Participants mark the line were appropriate between both extremes.
Sensory properties and palatability of the test meal after ingestion | Immediately following test meal ingestion (single measure)
  Participants will rate each test meal on their perceived sensory properties and rate different aspects related to its palatability. These are important considerations when developing new products and will be assessed using the validated visual analogue scale (VAS) method. The Visual Analogue Scale is a 100mm scale with anchors on each end describing extreme answers. On the left side of the scale is the extreme negative response and the right side the positive response. Participants mark the line were appropriate between both extremes.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Roche, Prof, Principal Investigator — University College Dublin; Katy Horner, Dr, Principal Investigator — University College Dublin; Dominique Dardevet, Dr, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (INRAE); Giuseppe De Vito, Prof, Principal Investigator — University of Padua Department of Biomedical Science, Neuromuscular Physiology Laboratory
Locations (2):
- University college Dublin, Dublin, Leinster, Ireland
- University of Padua Department of Biomedical Science, Neuromuscular Physiology Laboratory, Padua, Italy

IPD SHARING:
Plan to Share IPD: No